CLINICAL TRIAL: NCT03804177
Title: The Effect Of Hyaluronic Acid And Melatonin With Systemic Administration of Vitamin C On Implant Stability After Immediate Implant Placement in Anterior and Premolar Region in Systemically Healthy Patients
Brief Title: The Effect Of Hyaluronic Acid And Melatonin With Systemic Administration of Vitamin C On Implant Stability After Immediate Implant in Anterior Region
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Nabil Abdelfatiah, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio25111987
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Immediate Dental Implant
Keywords: immediate implant; hyaluronic acid; melatonin; vitamin C

STUDY DESIGN:
Intervention Model Description: it is randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implant with hyaluronic melatonin vit c (Experimental): implant placement with topical application of hyaluronic and melatonin and systemic administration of vitamin C
  Interventions: Procedure: immediate implant placement with melatonin hyaluronic acid vit C
- immediate implant (Active Comparator): immediate implant placement alone without melatonin or hyauronic acid nor vitamin c
  Interventions: Procedure: immediate implant placement without melatonin hyaluronic acid vit C

INTERVENTIONS:
Procedure: immediate implant placement with melatonin hyaluronic acid vit C — immediate implant placement with melatonin and hyaluronic acid and systemic administration vitamin C
  Other Names: early implant placement
  Arms: implant with hyaluronic melatonin vit c
Procedure: immediate implant placement without melatonin hyaluronic acid vit C — immediate implant placement without melatonin and hyaluronic acid and systemic administration vitamin C
  Other Names: early implant placement
  Arms: immediate implant

SUMMARY:
The concept of immediate implant placement at the time of tooth extraction was first introduced by Schulte et al. on animal studies. Since then, many follow-up studies examining different variables have supported the concept of immediate implant placement. pioneered a major contribution to immediate implant placement in human studies which recommended the insertion of an implant into a fresh extraction socket.

They advocated immediate implant placement primarily to reduce the number of surgical interventions needed to perform an implant-supported rehabilitation and shorten the treatment time.

Placement of implants immediately into extraction sites allow the surgeon to idealize the position of the implant appropriately with a better rehabilitation of the normal contour to the facial aspect of the final restoration.

Immediate implant placement in fresh extraction sockets was reported to reduce alveolar bone resorption. Better esthetic outcomes were achieved including the prosthetic crown length in harmony with the adjacent teeth, natural scalloping and easier distinct papillae to achieve and maximum soft tissue support.

Hyaluronic acid is a glycosaminoglycan, this unique molecule is implicated In a variety of biological functions including structural integrity, and the regulation of embryologic development. It is described as a natural organic substance, with physiological therapy activity, main component of the extracellular matrix of many tissues such as the skin, synovial joints and periodontal tissues .

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60.
2. Systemically healthy patients indicated for single or multiple immediate implants in anterior and premolar region.
3. Absence of any peri-apical pathosis.
4. Patients with intact buccal plate of bone.
5. Patients with adequate bone volume for the dental implant procedure.
6. Patient consent approval and signing.

Exclusion Criteria:

* 1. Smokers. 2. Systemic disease that may affect the final outcome of the surgical procedure.

  3. No or poor patient's compliance. 4. Patients with psychological problems. 5. Pathology at the site of intervention. 6. Pregnant patients. 7. Patients refuse to sign an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-02-10 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
implant stability | 6 months
  implant stability by ostell

SECONDARY OUTCOMES:
soft tissue healing | 6 months
  soft tissue healing by likert scale (0 indicate complete soft tissue Closure (no line of fibrin) , 1 indicate complete closure (thin line of fibrin) , 2 indcate complete closure (fibrin) , 3 indicate in complete closure (dehiscence ) , 4 indicate incomplete closure (necrosis)

CONTACTS AND LOCATIONS:
Overall Officials: Mona darhous, PHD, Study Chair — Cairo University; Mona shoieb, PHD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
i will check with my study chair

REFERENCES:
- [Background] Lee JH, Kim J, Baek HR, Lee KM, Seo JH, Lee HK, Lee AY, Zheng GB, Chang BS, Lee CK. Fabrication of an rhBMP-2 loaded porous beta-TCP microsphere-hyaluronic acid-based powder gel composite and evaluation of implant osseointegration. J Mater Sci Mater Med. 2014 Sep;25(9):2141-51. doi: 10.1007/s10856-014-5250-0. Epub 2014 Jun 14. PMID 24928668
- [Background] El-Gammal MY, Salem AS, Anees MM, Tawfik MA. Clinical and Radiographic Evaluation of Immediate Loaded Dental Implants With Local Application of Melatonin: A Preliminary Randomized Controlled Clinical Trial. J Oral Implantol. 2016 Apr;42(2):119-25. doi: 10.1563/aaid-joi-D-14-00277. Epub 2015 Jun 23. PMID 26103559